CLINICAL TRIAL: NCT02937181
Title: Antibiotic Prophylaxis With Ceftaroline for Type II and II Open Fractures: a Phase 4, Open-label, Prospective Clinical Trial
Brief Title: Antibiotic Prophylaxis in Open Fractures
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Olayemi Osiyemi MD (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Sponsor-Investigator, Olayemi Osiyemi MD, President/, Triple O Research Institute PA
Organization: Triple O Research Institute PA (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TEF-IT-40B
Record Dates: First submitted 2016-10-14; First posted 2016-10-18 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Open Fractures
MeSH Terms: conditions — Fractures, Open | interventions — Ceftaroline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- open fractures type II and III (Experimental): Every patients will receive Ceftaroline in an open label, single arm
  Interventions: Drug: Ceftaroline

INTERVENTIONS:
Drug: Ceftaroline — IV Ceftaroline will be given for 72 hours
  Other Names: Teflaro

SUMMARY:
Prospective look at antibiotic prophylaxis with Ceftaroline in patients with type II and III open fractures

DETAILED DESCRIPTION:
Determine if antibiotic prophylaxis with Ceftaroline in patients with type II and III open fractures is a safe and effective alternative to standard combination therapy

ELIGIBILITY:
Inclusion Criteria:

* male or female >= 18 years old
* complete an informed consent
* patients are diagnosed with a type II or III open fracture

Exclusion Criteria:

* allergy to beta-lactam antibiotics prior to screening
* prior to enrollment: patients received 3 or more doses of antibiotic prophylaxis
* pregnant female
* inability to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-12; Primary Completion 2018-10 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Rate of fracture site infection at 30 days between ceftaroline and historical hospital rate | 30 days

SECONDARY OUTCOMES:
Incidence of acute kidney injury | 30 days

OTHER OUTCOMES:
Identify bacteria associated with the infections | 30 days
identify the number of infections associated with sites other than fracture site | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Olayemi Osiyemi, MD, Principal Investigator — Triple O Research Institute PA
Locations (1):
- Triple O Research Institute PA, West Palm Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
no personal data, identifier and the data are made available